CLINICAL TRIAL: NCT06520631
Title: Response Of Arteriovenous Fistula Puncture-related Pain To Cryotherapy Application In Haemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Fathy Mohamed Elsaid, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005168
Record Dates: First submitted 2024-07-10; First posted 2024-07-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cryotherapy to arteriovenous fistula puncture site (Active Comparator): This group of patients receives ice pack applied on the site of the cannulation, for 20 sessions (3 sessions per week) it introduced for 5-10 minutes before the beginning of the dialysis.
  Interventions: Other: Ice packs (cryotherapy)
- Cryotherapy to site opposite to arteriovenous fistula puncture site (Active Comparator): This group of patients receives ice pack applied on contralateral to the site of the cannulation, for 20 sessions (3 sessions per week) it introduced for 5-10 minutes before the beginning of the dialysis.
  Interventions: Other: Ice packs (cryotherapy)

INTERVENTIONS:
Other: Ice packs (cryotherapy) — One group of patients receives ice pack applied on the site of the cannulation, for 20 sessions (3 sessions per week) it introduced for 5-10 minutes before the beginning of the dialysis.
  The second group of patients receives ice pack applied on contralateral to the site of the cannulation, for 20 sessions (3 sessions per week) it introduced for 5-10 minutes before the beginning of the dialysis.

SUMMARY:
Kidney disease occurs when kidney reduces its normal function, less than 30% of normal activity is related to a long-term condition. Therefore, people need to participate in a haemodialysis (HD) programme. In HD, blood is filtered by an external machine, done about three times a week and the access is gained through intermittent vascular cannulation.

The patients experience considerable pain due to the frequent insertion of AVF catheters.

Hemodialysis patients experience anxiety before needle insertion due to repeated punctures, and over 90% of patients experience acute pain during the process.

Puncture-related pain during arteriovenous fistula (AVF) cannulation in particular is a crucial influential factor in quality of life.

Cryotherapy is one of the interventions used in several studies to alleviate the arteriovenous fistula puncture-related pain. It can be conduct by using ice packs and the results of the previous studies have also shown its positive effects on the relief of the fistula puncture-related pain in these patients.

DETAILED DESCRIPTION:
Ninety male and female patients with end stage renal disease randomly assigned into three equal groups (n=30) their ages ranged between 30-50:

1. Group A (30 patients) receives ice pack applied on the site of the cannulation, for 20 sessions (3 sessions per week) it introduced for 5-10 minutes before the beginning of the dialysis.
2. Group B (30 patients) receives ice pack applied on contralateral to the site of the cannulation, for 20 sessions (3 sessions per week) it introduced for 5-10 minutes before the beginning of the dialysis.
3. Group C (30 patients) it is a control group this group not received ice pack.

ELIGIBILITY:
Inclusion Criteria:

* The study includes patients with ages from 30 to 50 years.
* Patients able to report pain adequately.
* Patients with end-stage kidney failure undergoing regular hemodialysis who have been treated for more than 3 months, at least twice per week, with arteriovenous fistula in use for more than 1 month are included in the study.

Exclusion Criteria:

Patients with conditions such as

* advanced age,
* advanced diabetes,
* cardiovascular insufficiency,
* cold allergy,
* Reynaud's phenomenon,
* nerve and tissue damage,
* fractures,
* heart failure,
* uncooperative patients,
* cognitive impairment preventing a proper assessment of pain.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2024-08-24 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS): | Visual analogue scale measured at baseline, and it will be measured again immediately after 20 sessions
  Scale to measure the intensity of pain The minimum value is 0 which means no pain and the maximum value is 10 which means the maximum pain

SECONDARY OUTCOMES:
The Arm Motor Ability Test (AMAT) | The Arm Motor Ability Test (AMAT): it is measured at baseline, and it will be measured again immediately after 20 sessions.
  The Arm Motor Ability Test (AMAT): is used to assess and quantify upper extremity functional limitation.
Hospital Anxiety and Depression Scale (HADS): | Hospital Anxiety and Depression Scale (HADS): it is measured at baseline, and it will be measured again immediately after 20 sessions.
  Hospital Anxiety and Depression Scale (HADS):
  it is a reliable and valid tool It's questions are clear and easy to understand, and thought the questionnaire items covered all patients problem areas regarding their hospital anxiety and depression. Each question is scored between 0 (no impairment) and 3 (severe impairment), with a maximum score of 21 means maximum impairment and minimum score of 0 means no impairment for anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Mohamed Badr, Professor, Study Director — Cairo University; Sahier Omar El-khashab, Professor, Study Director — Cairo university El-kasr el-aini
Locations (1):
- Cairo university, Cairo, Egypt